CLINICAL TRIAL: NCT07210307
Title: Forxiga (Dapagliflozin) Regulatory Post Marketing Surveillance
Brief Title: Safety Of DAPAGLIFLOZIN (FORXIGA) in Patient With Type 2 Diabetes Mellitus (T2dm) In Vietnam From A Post-Marketing Surveillance Program
Acronym: DAPAPMS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00038
Record Dates: First submitted 2025-05-21; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Safety Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is conducted to meet the requirements of the Drug Administration of Vietnam (DAV) on conducting necessary safety evaluations in routine clinical practice for a new medication within 3 years from its date of approval. For the case of the study treatment (dapagliflozin - Forxiga), safety and drug utilization reports have been regularly submitted by AstraZeneca to DAV every 6 months since its date of approval on 25th May 2016. To provide additional evidence on the safety profile of dapagliflozin in real-life settings and support renewing marketing authorizations for Forxiga, AstraZeneca collaborated with eight hospitals across Vietnam to implement this study.

DETAILED DESCRIPTION:
This study is a longitudinal observation on a cohort of 1001 patients with type 2 diabetes mellitus (T2DM), newly treated with dapagliflozin at eight hospitals across Vietnam. Adult T2DM patients who were newly treated with dapagliflozin and signed the informed consent form were eligibly recruited. For each recruited subject, the maximum duration of observation was 24 weeks, divided into 4 visits. In the first visit, data on subjects' baseline characteristics was collected. In the later visits, the presence, and the patterns of adverse events during the time treated with dapagliflozin were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* Diagnosed with T2DM, and eligible for initiating treatment with dapagliflozin according to indications of the approved summary of product characteristics of Forxiga in Vietnam.
* Provision of signed and dated written informed consent form by the potential study subject or the subject's legal guardian to demonstrate that s/he was informed necessary information of this study, prior to any mandatory study specific procedures

Exclusion Criteria:

* Patients who were prescribed dapaglifozin for off-label use (not mentioned in the approved summary of product characteristics of Forxiga in Vietnam)
* Patients who had contraindications with Forxiga

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort of interest included 1001 adult patients with T2DM who were newly treated with dapagliflozin (Forxiga). The sample size was determined in compliance with Vietnamese Ministry of Health's guidelines on conducting phase 4 clinical research to assess clinical benefits and risks of a medicinal product in real-life settings (8). According to this guideline, the minimal sample size for such a study is 1000 subjects. To achieve this targeted sample size, the total study period was expectedly 3 years.
Sampling Method: Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Annual incidence rate and proportions of AE, SAE, and sAR within 24 weeks | 24 weeks
  Monitoring and reporting data on adverse events (AEs) and serious adverse events (SAEs) during the treatment with dapagliflozin was implemented consistently with routine care in each studied site. For the patients discontinued dapagliflozin before completing the standard follow-up period (24 weeks), data would be collected via phone calls or emails. Decisions of continuing or discontinuing dapagliflozin treatment, either related or unrelated with safety issues, were completely depended on the medical doctor's opinion, with the patient's agreement

CONTACTS AND LOCATIONS:
Locations (1):
- HCMC Heart Institute, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690R00038&attachmentIdentifier=5551b81d-6e0a-4b1d-a17e-79b60f320ce7&fileName=D1690R00038_Redacted_CSR_Synopsis.pdf&versionIdentifier=